CLINICAL TRIAL: NCT01989247
Title: Self-management of Depression and Anxiety. A Randomized Controlled Trial.
Brief Title: How to Cope With Anxiety and Depression. A Randomized Controlled Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: National Board of Health, Denmark (Other Government); Danish Committee for Health Education (Other)
Responsible Party: Principal Investigator, Søren Christensen, Senior Researcher, University of Aarhus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-1010-46/1
Record Dates: First submitted 2013-11-14; First posted 2013-11-20 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Depression; Anxiety; Self Efficacy
Keywords: Depression; Anxiety; Randomized Controlled Trial; Self Care; Intervention Studies; Health Education
MeSH Terms: conditions — Depression; Anxiety Disorders; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-management program (Experimental): Seven weekly sessions of a group-based self-management programme for people with anxiety and depressive symptoms
  Interventions: Behavioral: Self-management programme
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Self-management programme — Seven weekly group-based sessions for people with anxiety and depressive symptoms
  Arms: Self-management program

SUMMARY:
The purpose of this study is to investigate whether citizens experiencing symptoms of anxiety and depression will benefit from a self-management training program with respect to: 1) Self-efficacy, and 2) Symptoms of anxiety and depression, and 3) Self reported measures of Health Related Quality of Life (HRQoL)

DETAILED DESCRIPTION:
* The intervention is a Danish adaption of The Chronic Disease Self-Management Program developed by The Stanford Patient Education Research Center, The Expert Patient Program Community Interest Company (EPPCIC), and The English National Health Service (NHS).
* The Danish adaptation has been performed by The Danish Committee for Health Education.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* Suffering from anxiety and/or depressive symptoms
* Voluntary participation

Exclusion Criteria:

* Potential suicidal behavior
* Potential aggressive behavior
* Significant cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 853 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Depressive Symptoms (Beck's Depression Inventory (BDI-II)) | Change from 1) Pre-randomization, to 2) Three months post-intervention
State Anxiety (Spielbergers State-Trait Anxiety Inventory (STAI)) | Change from 1) Pre-randomization, to 2) Three months post-intervention
  Only the State-anxiety subscale of the STAI is used
Self-efficacy (Chronic Disease Self-efficacy Scales - SECD-32 (Stanford Patient Education Research Center)) | Change from 1) Pre-randomization, to 2) Three months post-intervention
  Only the following subscale is used: "Obtain help from Community, Family, Friends Scale"
Self-efficacy ("Personal control" from "The Revised Illness Perception Questionnaire" (IPQ-R)) | Change from 1) Pre-randomization, to 2) Three months post-intervention
  Only the following subscale from the IPQ-R is used: "Personal Control"

SECONDARY OUTCOMES:
Sleep Quality (The Pittsburgh Sleep Quality Index) | Change from 1) Pre-randomization, to 2) Three months post-intervention
Exercise Behaviors (Stanford Patient Education Research Center) | Change from 1) Pre-randomization, to 2) Three months post-intervention
Health related symptoms | Change from 1) Pre-randomization, to 2) Three months post-intervention
  Self related overall health: Stanford Patient Education Research Center (1 item).
  Fatigue: Visual Analogue Scale. Stanford Patient Education Research Center (1 Item).
  Pain: Visual Analogue Scale. Stanford Patient Education Research Center (1 item).
Social/Role Activities Limitations Scale (Stanford Patient Education Research Center) | Change from 1) Pre-randomization, to 2) Three months post-intervention
Self-efficacy ("Control/Manage Depression Scale from: "Chronic Disease Self-efficacy Scales - SECD-32 (Stanford Patient Education Research Center)) | Change from 1) Pre-randomization, to 2) Three months post-intervention

OTHER OUTCOMES:
Common Mental Disorder Questionaire (CMDQ) | Change from 1) Pre-randomization, to 2) Three months post-intervention
  The following subscales are included: Somatization SCL-SOM; SCL-ANX4; SCL-DEP6; SCL-8
Well-being (WHO-5 Well Being Index) | Change from 1) Pre-randomization, to 2) Three months post-intervention
Coping (The Brief Cope) | Change from: 1) Pre-randomization, to 2) Three months post-intervention
Health Care Utilization | Change from 1) Pre-randomization, to 2) Three months post-intervention
  First two items from "Health Care Utilization" (Stanford Patient Education Research Center). Measured within the recent two months instead of six as used in the original scale.
Social Constraints (lepore) | Change from 1) Pre-randomization, to 2) Three months post-intervention
  Only the subscale refering to an "important other" was administered
Use of Health benefits | Change from 1) The full year prior to start of intervention, to 2) The three months period following the intervention
  Data on health benefits will be obtained by a linkage with The Danish National Health Insurance Service Registry

CONTACTS AND LOCATIONS:
Overall Officials: Soren Christensen, MSc, Principal Investigator — Aarhus University Hospital; Mimi Y Mehlsen, PhD, Study Director — University of Aarhus
Locations (37):
- Denmark (37):
  - Aalborg Municipality, Aalborg
  - Nordfyn Municipality, Bogense
  - Ikast-Brande Municipality, Brande
  - Gentofte Municipality, Charlottenlund
  - Dragør Municipality, Dragør
  - Helsingør Municipality, Elsinore
  - Esbjerg Municipality, Esbjerg
  - Vesthimmerlands Municipality, Farsø
  - Fredericia Municipality, Fredericia
  - Frederikssund Municipality, Frederikssund
  - Norddjurs Municipality, Grenå
  - Haderslev Municipality, Haderslev
  - Faxe Municipality, Haslev
  - Herning Municipality, Herning
  - Holbæk Municipality, Holbæk
  - Tårnby Municipality, Kastrup
  - Fredensborg Municipality, Kokkedal
  - Lyngby-Taarbæk Municipality, Kongens Lyngby
  - Køge Municipality, Køge
  - Hedensted Municipality, Løsning
  - Næstved Municipality, Næstved
  - Odense Municipality, Odense
  - Roskilde Municipality, Roskilde
  - Aabenraa Municipality, Rødekro
  - Syddjurs Municipality, Rønde
  - Silkeborg Municipality, Silkeborg
  - Skanderborg Municipality, Skanderborg
  - Slagelse Municipality, Slagelse
  - Solrød Municipality, Solrød Strand
  - Sorø Municipality, Sorø
  - Rebild Municipality, Støvring
  - Gladsaxe Municipality, Søborg
  - Sønderborg Municipality, Sønderborg
  - Varde Municipality, Varde
  - Vejen Municipality, Vejen Municipality
  - Vejle Municipality, Vejle
  - Viborg Municipality, Viborg